CLINICAL TRIAL: NCT00305422
Title: Efficacy of Quetiapine Compared to Risperidone on Negative Symptoms and Cognition With Regard to Underlying Neurobiological Mechanisms and Brain Activation.
Brief Title: Effect of Quetiapine on Negative Symptoms and Cognition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5077/9007
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate; Risperidone

INTERVENTIONS:
Drug: Quetiapine fumarate
Drug: Risperidone

SUMMARY:
The purpose of the study is to investigate the outcome on negative symptoms of schizophrenic patients during therapy with quetiapine or risperidone.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* men and women aged 18 to 65 years with diagnosis of schizophrenia
* score of at least 4 CGI, PANSS negative subscale score > 21
* fulfil the criterion to be right-handed for inclusion in the fMRI investigations

Exclusion Criteria:

* Substance or alcohol dependence
* female patients who are pregnant, lactating or at risk of pregnancy
* history of organic CNS-trauma, epilepsy, meningoencephalitis, psychosurgery, instable somatic conditions
* risk of suicide or aggressive behaviour
* history of electroconvulsive therapy, Parkinson's disease, Prolactin-dependent tumor

For the subset of subjects for the fMRI investigations the following additional exclusion criteria is valid as:

* existence of metal in the body as by cardiac pacemaker, coil, total prosthesis, metal splinter, metal articulation, metal balls.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2001-11; Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy of both neuroleptics, especially with regard to cognitive deficits and functional brain activation between baseline and week 12

SECONDARY OUTCOMES:
Change from baseline in PANSS negative symptom total score, PANSS subscores, CGI, CGI-severity of illness, HAMD, Simpson-Angus-Scale, BPRS, specific PANSS items , Startle reflex.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Germany Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Munich, Germany